CLINICAL TRIAL: NCT05623033
Title: The Predictive Value of Dynamic Changes of CD4+T Lymphocytes in Primary Nephrotic Syndrome With Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Guangdong traditional Chinese medicine hospital, Zhuhai (Unknown)
Responsible Party: Sponsor
Other Study IDs: WPZhu
Record Dates: First submitted 2022-11-07; First posted 2022-11-21 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Nephrotic Syndrome; Infections; Lymphocyte
MeSH Terms: conditions — Nephrotic Syndrome; Infections | interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infection group
  Interventions: Other: The study is an observational study without intervention
- non-infection group
  Interventions: Other: The study is an observational study without intervention

INTERVENTIONS:
Other: The study is an observational study without intervention — The study is an observational study without intervention

SUMMARY:
The goal of this observational study is to test whether the dynamic changes of CD4+T lymphocytes can predict infections in patients with primary nephrotic syndrome . The main questions it aims to answer are:

* whether the dynamic changes of CD4+T lymphocytes can predict infections in patients with primary nephrotic syndrome
* effect of different immunosuppressive therapy on the number and function of T lymphocyte subsets in patients with primary nephrotic syndrome

Participants will be divided into infection group and non-infection group according to whether they are infected

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 14 years and<75 years.
2. It meets the diagnostic criteria of primary nephrotic syndrome, i.e. a. A large amount of proteinuria (24h urine protein quantity > 3.5g/d); b. Hypoalbuminemia (liver function: albumin<30g/L); c. Edema; d. The blood lipid is elevated. Among them, item a and b are necessary conditions for diagnosis.
3. Nephrocentesis pathology indicates the pathological type of nephrotic syndrome (minimal change glomerulonephritis, membranous nephropathy, focal segmental glomerulonephritis, membranous proliferative glomerulonephritis, mesangial proliferative glomerulonephritis).
4. Glucocorticoids or corticosteroids combined with immunosuppressants should be used clinically.

Exclusion Criteria:

1. Secondary nephrotic syndrome, such as secondary to systemic lupus erythematosus, hepatitis B, hepatitis C, tumor, organic solvent , heavy metal poisoning, etc.
2. Patients with tumor and chronic infectious diseases, such as HIV infection, cardiac insufficiency, acute hepatitis, transaminase increase more than twice the normal value, deep vein thrombosis.
3. The subjects were pregnant and lactating women.
4. Patients with serious primary diseases such as heart, brain, liver and hematopoietic system.
5. Those who can not cooperate, such as the mentally ill.
6. It is known that it is allergic to or has contraindications to any component in glucocorticoid, FK506, MMF and CTX.
7. Serum creatinine (SCR) > 265.2 μ mol/L（3mg/dl）。

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with primary nephrotic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2022-11-16 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dynamic changes of CD4+T cells | 3 years after the project starts
  Whether the change of CD4+T lymphocytes count can predict infections in patients with primary nephrotic syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- the fifth affiliated hospital of SUN YAT-SEN university, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No